CLINICAL TRIAL: NCT00335010
Title: A Prospective Double Blinded Study on the Effect of Intravenously Administrated Nitroglycerine on Gastric Tissue Microvascular Bloodflow and Microvascular Hemoglobin Saturation During Gastric Tube Reconstruction
Brief Title: Intravenous NTG to Preserve Gastric Microcirculation During Gastric Tube Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MEC-2004-160
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2006-06-08 (Estimated); Status verified 2006-06

CONDITIONS: Esophageal Neoplasms; Microcirculation
Keywords: Nitroglycerine; gastroesophageal anastomosis; microvascular bloodflow; microvascular hemoglobinsaturation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin

SUMMARY:
The aim of the present study was to investigate if NTG, administered intravenously during gastric tube reconstruction, could preserve gastric fundus tissue blood flow and oxygenation and reduce the incidence of postoperative leakage.

DETAILED DESCRIPTION:
Complications of oesophagectomy and gastric tube reconstruction are leakage and stenosis, which may be due to compromised microvascular blood flow (MBF) in the gastric tissue. We recently demonstrated that peri-operatively decreased MBF could be improved by topical administration of nitro-glycerine NTG). In this present study we investigate the effect of intravenous NTG on gastric microcirculation.

This single centre, prospective, double blinded study randomized thirty-two patients scheduled for esophagectomy into two groups. The intervention group received intravenous NTG during gastric tube reconstruction, as the control group received normal saline.

Baseline values of MBF, microvascular haemoglobin O2 saturation (μHbSO2), and microvascular haemoglobin concentration (μHbcon) were determined at the gastric fundus before and after gastric tube construction and after pulling up the gastric tube to the neck.

ELIGIBILITY:
Inclusion Criteria:

* Planned esophagectomy with gastric tube reconstruction
* written informed consent
* ASA I and II

Exclusion Criteria:

* younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2005-05; Study Completion 2005-12

PRIMARY OUTCOMES:
differences in Microvascular bloodflow
differences in microvascular hemoglobinsaturation

SECONDARY OUTCOMES:
differences in anastomotic leakage
differences in anastomotic stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Gommers, MD, PhD, Study Chair — Erasmus Medical Center; Marc Buise, MD, Principal Investigator — Erasmus Medical Center; Jasper van Bommel, MD, PhD, Study Director — Erasmus Medical Center; Huug Tilanus, MD, PhD, Principal Investigator — Erasmus Medical Center; Khe Tran, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Background] Buise MP, Ince C, Tilanus HW, Klein J, Gommers D, van Bommel J. The effect of nitroglycerin on microvascular perfusion and oxygenation during gastric tube reconstruction. Anesth Analg. 2005 Apr;100(4):1107-1111. doi: 10.1213/01.ANE.0000147665.60613.CA. PMID 15781529
- [Background] Pierie JP, de Graaf PW, van Vroonhoven TJ, Obertop H. Healing of the cervical esophagogastrostomy. J Am Coll Surg. 1999 Apr;188(4):448-54. doi: 10.1016/s1072-7515(99)00003-4. No abstract available. PMID 10195730
- [Background] Jacobi CA, Zieren HU, Zieren J, Muller JM. Is tissue oxygen tension during esophagectomy a predictor of esophagogastric anastomotic healing? J Surg Res. 1998 Feb 1;74(2):161-4. doi: 10.1006/jsre.1997.5239. PMID 9587355
- [Background] Siegemund M, van Bommel J, Ince C. Assessment of regional tissue oxygenation. Intensive Care Med. 1999 Oct;25(10):1044-60. doi: 10.1007/s001340051011. No abstract available. PMID 10551958
- [Derived] Buise M, van Bommel J, Jahn A, Tran K, Tilanus H, Gommers D. Intravenous nitroglycerin does not preserve gastric microcirculation during gastric tube reconstruction: a randomized controlled trial. Crit Care. 2006;10(5):R131. doi: 10.1186/cc5043. PMID 16970804